CLINICAL TRIAL: NCT05156684
Title: Evaluating the Therapeutic Effect of Pentoxifylline and Zinc Co-administration in Patients With Idiopathic Oligoasthenoteratozoospermia
Brief Title: Effect of Pentoxifylline and Zinc Co-administration in Patients With Oligoasthenoteratozoospermia
Acronym: OAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Arak University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zeynab, Principal Investigator, Arak University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 96/197
Record Dates: First submitted 2021-11-05; First posted 2021-12-14 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Idiopathic Infertility
MeSH Terms: interventions — Pentoxifylline; Zinc; Zinc Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- placebo group (Experimental): Control group: oral rehydration salts (ORS, Poursina, Tehran, Iran), two times daily
  Interventions: Drug: Placebo
- pentoxifylline group (Experimental): Intervention group 1: received pentoxifylline (TRENTAL 400 mg modified release tablets, OSPS; 400 mg ,two times daily)
  Interventions: Drug: Pentoxifylline
- Zinc group (Experimental): Intervention group 2: received zinc ( Zinc Sulfate 220mg Capsules,One time daily)
  Interventions: Drug: zinc
- pentoxifylline+ zinc group (Experimental): Intervention group 3: received pentoxifylline+ zinc (TRENTAL 400 mg modified release tablets, OSPS; 400 mg ,two times daily + Zinc Sulfate 220mg Capsules,One time daily )
  Interventions: Drug: zinc + pentoxifylline

INTERVENTIONS:
Drug: Placebo — Infertile men referred to the infertility treatment center who, have had at least one year of unprotected intercourse, Natural fertility has not happened in their spouse. These men will all be married These men will be between the ages of 20 and 50. According to WHO criteria, Sperm parameters abnormalities should be observed in at least two spermogram within 2 weeks. Candidates receive two placebo tablets daily
  Other Names: hydration solution
  Arms: placebo group
Drug: Pentoxifylline — Infertile men referred to the infertility treatment center who, have had at least one year of unprotected intercourse, Natural fertility has not happened in their spouse. These men will all be married These men will be between the ages of 20 and 50. According to WHO criteria, Sperm parameters abnormalities should be observed in at least two spermogram within 2 weeks. Candidates receive two trental tablets daily
  Other Names: Trental
  Arms: pentoxifylline group
Drug: zinc — Infertile men referred to the infertility treatment center who, have had at least one year of unprotected intercourse, Natural fertility has not happened in their spouse. These men will all be married These men will be between the ages of 20 and 50. According to WHO criteria, Sperm parameters abnormalities should be observed in at least two spermogram within 2 weeks. Candidates receive one zinc sulfate tablet daily
  Other Names: zinc sulfate
  Arms: Zinc group
Drug: zinc + pentoxifylline — Infertile men referred to the infertility treatment center who, have had at least one year of unprotected intercourse, Natural fertility has not happened in their spouse. These men will all be married These men will be between the ages of 20 and 50. According to WHO criteria, Sperm parameters abnormalities should be observed in at least two spermogram within 2 weeks. Candidates receive two pentoxifylline tablets+ one zinc tablet daily
  Other Names: zinc sulfate+ trental
  Arms: pentoxifylline+ zinc group

SUMMARY:
The aim of this study is to investigate the impact of co-administration of Pentoxifylline and Zinc sulfate on oxidative stress, apoptosis, and inflammation, sperm capacitation and parameters in infertile men.

DETAILED DESCRIPTION:
This study will be performed as a double-blind randomized clinical trial on idiopathic infertile men (including oligoasthenosospermia, dyspnea, astheno-teratozoospermia, oligo-astheno-teratozoospermia) referred to Shafa Infertility Clinic. Patient satisfaction, non-use of contraceptives, men aged 25 to 43 years and idiopathic infertility according to WHO criteria (World Health, 2010) are our study criteria. A food questionnaire is also taken from them to identify patients. Any medication that may affect sperm production should be discontinued within three months of the study.

Sampling and administration of pentoxifylline and zinc:

Preparation and analysis of semen samples are performed according to WHO 2010 recommendations. Semen samples are prepared by masturbating after a 3 to 5 day abstinence period. Two semen samples from these men, one before and the other after the intervention, are evaluated for basic parameters. For liquefaction, semen samples are incubated for 30 to 60 minutes at 37 ° C. Microscopic tests are performed to evaluate indicators such as sperm concentration in semen, motility and sperm morphology. Objectives and study methods are explained to patients who meet the inclusion criteria. Written consent is then obtained from the candidate. Body mass index (BMI) is assessed for patients. Also, at the beginning of the study, 5 cc of blood is taken from patients to measure reproductive hormones.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic infertile men
* have had at least one year of unprotected intercourse infertility
* Sperm parameters abnormality

Exclusion Criteria:

* Men with varicocele
* Hypersensitivity to pentoxifylline & zinc,
* pelvic organic pathologies
* congenital adrenal hyperplasia
* thyroid dysfunction
* Cushing's syndrome
* hyper prolactinemia
* androgen secreting neoplasia
* diabetes mellitus
* consumption of medications affecting carbohydrate metabolism
* severe hepatic
* pancreatitis
* kidney diseases
* gallbladder diseases
* Patients with alcohol consumption
* Patients who use cigarettes and drugs

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — men with idiopathic infertility
Enrollment: 140 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-01-10 (Estimated); Study Completion 2022-05-28 (Estimated)

PRIMARY OUTCOMES:
count of sperm | One week after starting the medication
  count of sperm(In per million - with the help of a neobar slide and microscopic observation
motility of sperm | One week after starting the medication
  motility of sperm: Calculate the percentage of motile sperm using microscopic observation
morphology of sperm | One week after starting the medication
  Calculate the percentage of sperm with a normal shape with the help of Papanic staining
Malon di aldehyd evaluate | One week after starting the medication
  Malondialdehyde (nmol/mL), will be measured using related experimental kits
ROS evaluate | One week after starting the medication
  reactive oxygen species (ROS (RLU/s)), will be measured using related experimental kits
TAC (Total Antioxidant Capacity) evaluate | One week after starting the medication
  total antioxidant capacity (TAC (/m / l)) will be measured using related experimental kits
FSH hormon | One week after starting the medication
  FSH (IU / L) will be measured from the blood serum of volunteers using ELISA kit
LH hormon | One week after starting the medication
  LH (IU / L) will be measured from the blood serum of volunteers using ELISA kit
Testosteron hormon | One week after starting the medication
  testosterone (nanomolar per liter) will be measured from the blood serum of volunteers using ELISA kit
TNF α( Tissue necrosis Factor) | One week after starting the medication
  TNF α( Tissue necrosis Factor) (pg/mL) as an inflammatory factor will be measured using related experimental kit
Interleukin-6 (IL-6) | One week after starting the medication
  Interleukin-6 (IL-6)/(pg/mL) as an inflammatory factor will be measured using related experimental kit
Sperm DNA Fragmentation Assay(SDFA) | One week after starting the medication
  DNA fragmentation will be assessed using an SDFA kit and microscopic observations (as a percentage of damaged sperm).

OTHER OUTCOMES:
caspase 3 expression | 3 months
  expression of caspase 3 gen (in p.c) using real-time PCR and Western blot
BAX expression | 3 months
  expression of BAX gen(in p.c) using real-time PCR and Western blot
BCL 2 expression | 3 months
  expression of BCL 2 gen (in p.c) using real-time PCR and Western blot

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dadgar Z, Shariatzadeh SMA, Mehranjani MS, Kheirolahi A. The therapeutic effect of co-administration of pentoxifylline and zinc in men with idiopathic infertility. Ir J Med Sci. 2023 Feb;192(1):431-439. doi: 10.1007/s11845-022-02931-0. Epub 2022 Feb 19. PMID 35182288